CLINICAL TRIAL: NCT01967004
Title: Validation of a Control Method for Upper Limb Myoelectric Prostheses Using Radio Frequency Identification (RFID)
Brief Title: Enhancing Upper Limb Prostheses With Radio Frequency Identification
Acronym: RFIDIBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Infinite Biomedical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RFID-IBT-3600
Record Dates: First submitted 2013-09-26; First posted 2013-10-22 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2013-10

CONDITIONS: Below Elbow Amputation

ARMS (1):
- Functional Assessment (Experimental): Participant will be asked to perform a series of tasks involving their prosthesis. These tasks can involve switching grips as well as moving objects.
  Interventions: Device: Morph

INTERVENTIONS:
Device: Morph — Morph is a small electric controller that is retrofit into existing myoelectric prostheses to equip them with wireless identification capabilities. Specifically, Morph allows the prosthesis to react to RFID tags in the environment.
  Other Names: Myoelectrically-Operated RFID Prosthetic Hand

SUMMARY:
The purpose of this study is to determine if Radio Frequency Identification (RFID) can lead to greater prosthesis function and control. Subjects are asked to perform specific tasks and actions using the traditional control method, as well as RFID control.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or greater.
2. Below elbow amputation, unilateral or bilateral.
3. Chronic stable amputation: > 6 months from amputation.
4. Stable prosthesis prescription: > 3 months since last major prosthesis modification.
5. Cognitively intact, as determined by Mini-Mental Status Examination score > 24.
6. Able to provide informed consent and available to participate in study activities.
7. No severe residual limb motor/sensory impairment or pain likely to interfere with treatment.
8. Expected to be medically and psychiatrically stable for study duration.

Exclusion Criteria:

1. Patients with diseases which weaken and/or adversely affect the control of skeletal muscle.
2. Patients with poor skin integrity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-04 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Time required to perform different functional tasks | 12 weeks
  Each participant will perform functional tests on the first visit. These tests consist of moving objects from one location to another, and performing certain muscle contraction patterns when prompted. The participant will then take the prosthesis, installed with morph, home for 3 months at most, and then return to perform another set of timed trials.

SECONDARY OUTCOMES:
Questionnaires on prosthesis function and satisfaction | 20 minutes per questionnaire, total of 3 different questionnaires administered twice each
  The questionnaires offer the participant the opportunity to express their experience and satisfaction with their prosthesis, during different tasks and at home.

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Eastern Campus, Baltimore, Maryland, United States